CLINICAL TRIAL: NCT04500353
Title: A Randomised Trial of Routine or Selective Application of a Face Mask for Preterm Infants at Birth
Brief Title: Routine Or Selective Application of a Face Mask for Preterm Infants at Birth: the ROSA Trial
Acronym: ROSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROSA.01
Record Dates: First submitted 2020-07-24; First posted 2020-08-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Infant, Premature, Diseases; Continuous Positive Airway Pressure; Positive-Pressure Respiration; Resuscitation; Respiratory Distress Syndrome, Newborn
MeSH Terms: conditions — Infant, Premature, Diseases; Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Intervention Model Description: Randomised parallel group study
Masking Description: Masking of caregivers not feasible due to the nature of the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine face mask application (Active Comparator): Routine application of a face mask shortly after birth to deliver continuous positive airway pressure (CPAP)
  Interventions: Other: Face mask application for CPAP and/or PPV delivery
- Selective face mask application (Experimental): Selective application of a face mask to give positive pressure ventilation (PPV) for apnoea or bradycardia [heart rate (HR) < 100 beats per minute (bpm)] at any time in the delivery room (DR); or to give CPAP for signs of respiratory distress after 5 minutes of life
  Interventions: Other: Face mask application for CPAP and/or PPV delivery

INTERVENTIONS:
Other: Face mask application for CPAP and/or PPV delivery — Face mask application for CPAP and/or PPV delivery

SUMMARY:
International guidelines recommend giving positive pressure ventilation (PPV) by face mask to newborns who do not breathe or have a slow heart rate at birth. Preterm infants are at high risk of developing respiratory distress syndrome (RDS) and many are treated with continuous positive airway pressure (CPAP) in the neonatal intensive care unit (NICU). Though the majority of preterm infants breathe spontaneously at birth, many clinicians routinely apply a face mask to preterm infants shortly after birth in the delivery room (DR) to give them CPAP. However, applying a face mask may inhibit spontaneous breathing in newborns. In this study, premature babies will be randomly assigned to have a face mask routinely applied for CPAP shortly after birth; or to have a face mask selectively applied only for PPV if they are not breathing or have a slow heart beat in the first 5 minutes of life, or for CPAP if they have signs of respiratory distress after 5 minutes. The investigators will determine whether fewer participants who have the mask selectively applied receive PPV in the DR.

DETAILED DESCRIPTION:
Newly born babies have fluid-filled lungs that they must quickly aerate after birth. Compared to infants born at term, preterm babies have greater difficulty in establishing and maintaining aeration of their lungs; this leaves them at increased risk of developing respiratory distress syndrome (RDS). Infants who develop RDS are treated with nasal continuous positive airway pressure (CPAP), and may progress to treatment with surfactant and mechanical ventilation, in the Neonatal Intensive Care Unit (NICU).

The Neonatal Task Force of the International Liaison Committee on Resuscitation (ILCOR) makes recommendations on the treatment of infants at birth. ILCOR recommends assessing the breathing and heart rate (HR) of all newborns, and:

1. Giving positive pressure ventilation (PPV) to babies who have a HR < 100bpm, gasping or apnoea
2. Considering giving CPAP to babies who have laboured breathing or persistent cyanosis

Most preterm infants breathe spontaneously at birth. Despite this, the majority of preterm infants have a facemask applied for respiratory support immediately after birth, usually before the HR has been determined. Clinicians presumably do this to give early support to infants they believe are at high risk of developing RDS in an attempt to prevent or lessen the severity of the disease.

There is little evidence that giving preterm infants prophylactic nasal CPAP may be superior to supportive care with oxygen. A study that compared nasopharyngeal CPAP to supportive care with oxygen performed before antenatal steroids were routinely given found no difference in the rate of development of RDS with the application of CPAP. Two more recent studies did not show that early application of nasal CPAP reduced the rate of intubation or treatment with surfactant. In these studies CPAP was given by nasal prongs and was started at 15 - 30 minutes of life, not immediately with a facemask. There is no evidence that facemask CPAP immediately after birth prevents or reduces the severity of RDS.

Application of a face mask has been demonstrated to inhibit spontaneous breathing in many term infants. Cold gas flow, such as that provided by a T-piece, can inhibit spontaneous breathing in term infants. Application of a face mask for breathing support appears to inhibit breathing in a greater proportion of preterm infants. Considerable force is applied to the head when face mask PPV is given to a mannequin in the supine position.

Routinely applying a face mask for respiratory support may be unnecessary in many premature babies. It may inhibit their spontaneous breathing and result in them receiving facemask PPV more frequently in the DR. It may also affect how well they breathe in the first day of life and increase the rate of treatment with nasal CPAP in the NICU.

METHODS

RANDOMISATION AND GROUP ASSIGNMENT Participants will be randomly assigned to "SELECTIVE" or "ROUTINE" groups in a 1:1 ratio. The group assignment schedule will be generated in blocks of 4 using a random number table, and will be stratified by gestational age (23 - 27, 28 - 31+6). It will be kept on a concealed from investigators and treating clinicians. Group assignment will be written on cards and placed in sequentially numbered, sealed, opaque envelopes. Infants of multiple gestations will be randomised as individuals.

The envelopes will be contained in 2 boxes for GA strata and kept in the NICU. The next envelope in the sequence will be taken from the appropriate box and brought to the DR, where it will be opened just before delivery.

MASKING It is not possible to mask caregivers to group assignment.

INTERVENTIONS

ALL INFANTS Infants in both groups will have their umbilical cord clamped at or after 1 minute of age; they will not have a mask applied for respiratory support during this time. Infants will then be transferred to resuscitaire, placed supine under radiant heat and have a hat applied. All infants will be placed in polyethylene bag. A pulse oximeter will be placed on the right wrist.

A T-piece device (Neopuff, Fisher & Paykel Healthcare, Auckland NZ; or Dräger Resuscitaire (Drager healthcare, Lübeck, Germany) and round face mask (Fisher & Paykel Healthcare, Auckland NZ) of appropriate size for the baby will be used to give respiratory support to infants in both groups. The T-piece will have gas flow set at 8 - 10 L/min, with settings PEEP 6cmH2O, and PIP 25cmH2O. There will be an air/oxygen blender in the circuit and the FiO2 will be initially set at 30%. The FiO2 will not be adjusted before 5 minutes of age.

SELECTIVE GROUP Infants assigned to the "SELECTIVE" group will be placed supine to breathe spontaneously. If SpO2 < 70% at 5 minutes and their respiratory effort is good, they will be given give free flow oxygen (i.e. the mask will be placed in front of, but not directly in contact with, the infant's face). The FiO2 may be increased at 1 minute intervals thereafter, aiming for SpO2 ≥ 90% at 10 minutes of life.

Infants in the "SELECTIVE" group will have mask PPV if they are apnoeic or have HR < 100bpm at any time in the DR. Clinicians may consider applying facemask to give CPAP if the infants breathing is laboured (i.e. there are signs of respiratory distress - grunting, intercostal/subcostal/sternal recessions) after 5 minutes of age.

ROUTINE GROUP Infants assigned to the "ROUTINE" group will be placed supine on the resuscitaire and have facemask CPAP applied as soon as possible after they arrive. If SpO2 < 70% at 5 minutes, the FiO2 may be increased at 1 minute intervals, aiming for SpO2 ≥ 90% at 10 minutes of life.

Infants in the "ROUTINE" group will have facemask PPV if they are apnoeic or have HR < 100bpm at any time in the DR. Mask respiratory support may be withdrawn as and when desired by clinical staff.

RESUCE TREATMENT All other treatments - i.e. endotracheal intubation for PPV, chest compressions, adrenaline, volume - w ill be given at the discretion of the treating clinicians and in accordance with ILCOR recommendations.

SAMPLE SIZE ESTIMATION To show a reduction in the proportion of babies receiving PPV with routine application from 60% to 40% with selective application with 80% power and α of 0.05, the investigators need to recruit 200 infants.

ELIGIBILITY:
Inclusion Criteria:

* Born before 32 weeks gestational age by best obstetric estimate

Exclusion Criteria:

* Infants with major congenital anomalies

Ages: 0 Minutes to 5 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 201 (Actual)
Dates: Start 2020-10-11 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
The proportion of participants who receive face mask PPV in the delivery room DR | Within 30 minutes of birth
  The proportion of participants who receive face mask positive pressure ventilation (PPV) in the delivery room (DR)

SECONDARY OUTCOMES:
The proportion of participants who receive face mask CPAP in the first 5 minutes of life | 5 minutes
  The proportion of participants who receive face mask (continuous positive airway pressure) CPAP in the first 5 minutes of life
The proportion of participants who receive face mask PPV in the first 5 minutes of life | 5 minutes
  The proportion of participants who receive face mask PPV in the first 5 minutes of life
HR at 5 minutes of life | 5 minutes
  Heart rate (HR) at 5 minutes of life
SpO2 at 5 minutes of life | 5 minutes
  Oxygen saturation (SpO2) at 5 minutes of life
The proportion of participants who receive face mask CPAP in the DR | Within 30 minutes of birth
  The proportion of participants who receive face mask CPAP in the DR
Duration of PPV in the DR | Within 30 minutes of birth
  Duration of PPV in the DR
The proportion of participants who are intubated in the DR | Within 30 minutes of birth
  The proportion of participants who are intubated in the DR
The proportion of participants who receive chest compressions in the DR | Within 30 minutes of birth
  The proportion of participants who receive chest compressions in the DR
The proportion of participants who receive volume in the DR | Within 30 minutes of birth
  The proportion of participants who receive volume in the DR
The proportion of participants who receive adrenaline in the DR | Within 30 minutes of birth
  The proportion of participants who receive adrenaline in the DR
Maximum FiO2 in the DR | Within 20 minutes of birth
  Maximum fraction of inspired oxygen (FiO2) in the DR
Apgar score at 5 minutes | 5 minutes
  Apgar score at 5 minutes (scale 0 -10, higher scores indicate better outcome)
Apgar score at 10 minutes | 10 minutes
  Apgar score at 10 minutes (scale 0 -10, higher scores indicate better outcome)
Respiratory support in transport to NICU | Within 45 minutes of birth
  Respiratory support in transport to the neonatal intensive care unit (NICU)
The proportion of participants who receive NCPAP in NICU | Within one month
  The proportion of participants who receive nasal CPAP in NICU
The proportion of participants who receive endotracheal ventilation in NICU | Within one month
  The proportion of participants who receive endotracheal ventilation in NICU
The proportion of participants who receive surfactant treatment | Within one month
  The proportion of participants who receive surfactant treatment
The proportion of participants who have a pneumothorax drained | Within one month
  The proportion of participants who have a pneumothorax drained
The proportion of participants who survive free of BPD | Day 28 of life
  The proportion of participants who are alive and not receiving respiratory support or supplemental oxygen on day 28 of life
The proportion of participants who receive survive free of CLD | 36 weeks corrected
  The proportion of participants who are alive and not receiving respiratory support or supplemental oxygen at 36 weeks corrected age
The proportion of participants who receive postnatal steroids | Through study completion, an average of 2-3 months in survivors
  The proportion of participants who receive postnatal steroids
The proportion of participants who receive home oxygen therapy | Through study completion, an average of 2-3 months in survivors
  The proportion of participants who receive home oxygen therapy
The proportion of participants who die before hospital discharge | Through study completion, an average of 2-3 months in survivors
  The proportion of participants who die before hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Colm PF O'Donnell, PhD, Principal Investigator — National Maternity Hospital; University College Dublin
Locations (1):
- National Maternity Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be shared for studies approved by the chief and principal investigators
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available after the primary report of the study has been published and will be available for 5 years
Access Criteria: Requests for data that are accompanied by a protocol that describes the nature and purpose of the study, the data that is required and how it will be analysed will be considered by the chief and principal investigators. Studies that are determined not to be contrary to partcipants' interests; and to be consistent with the purpose for which consent was given for the original study and methodologically sound may be approved

REFERENCES:
- [Background] Perlman JM, Wyllie J, Kattwinkel J, Wyckoff MH, Aziz K, Guinsburg R, Kim HS, Liley HG, Mildenhall L, Simon WM, Szyld E, Tamura M, Velaphi S; Neonatal Resuscitation Chapter Collaborators. Part 7: Neonatal Resuscitation: 2015 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2015 Oct 20;132(16 Suppl 1):S204-41. doi: 10.1161/CIR.0000000000000276. No abstract available. PMID 26472855
- [Background] O'Donnell CP, Kamlin CO, Davis PG, Morley CJ. Crying and breathing by extremely preterm infants immediately after birth. J Pediatr. 2010 May;156(5):846-7. doi: 10.1016/j.jpeds.2010.01.007. Epub 2010 Mar 16. PMID 20236659
- [Background] Murphy MC, McCarthy LK, O'Donnell CPF. Crying and breathing by new-born preterm infants after early or delayed cord clamping. Arch Dis Child Fetal Neonatal Ed. 2020 May;105(3):331-333. doi: 10.1136/archdischild-2018-316592. Epub 2019 May 13. PMID 31085675
- [Background] Katheria A, Arnell K, Brown M, Hassen K, Maldonado M, Rich W, Finer N. A pilot randomized controlled trial of EKG for neonatal resuscitation. PLoS One. 2017 Nov 3;12(11):e0187730. doi: 10.1371/journal.pone.0187730. eCollection 2017. PMID 29099872
- [Background] Kuypers KLAM, Lamberska T, Martherus T, Dekker J, Bohringer S, Hooper SB, Plavka R, Te Pas AB. The effect of a face mask for respiratory support on breathing in preterm infants at birth. Resuscitation. 2019 Nov;144:178-184. doi: 10.1016/j.resuscitation.2019.08.043. Epub 2019 Sep 12. PMID 31521774
- [Background] Murphy MC, McCarthy LK, O'Donnell CPF. Initiation of respiratory support for extremely preterm infants at birth. Arch Dis Child Fetal Neonatal Ed. 2021 Mar;106(2):208-210. doi: 10.1136/archdischild-2020-319798. Epub 2020 Aug 26. PMID 32847832
- [Background] Subramaniam P, Ho JJ, Davis PG. Prophylactic nasal continuous positive airway pressure for preventing morbidity and mortality in very preterm infants. Cochrane Database Syst Rev. 2016 Jun 14;(6):CD001243. doi: 10.1002/14651858.CD001243.pub3. PMID 27315509
- [Background] Sandri F, Ancora G, Lanzoni A, Tagliabue P, Colnaghi M, Ventura ML, Rinaldi M, Mondello I, Gancia P, Salvioli GP, Orzalesi M, Mosca F. Prophylactic nasal continuous positive airways pressure in newborns of 28-31 weeks gestation: multicentre randomised controlled clinical trial. Arch Dis Child Fetal Neonatal Ed. 2004 Sep;89(5):F394-8. doi: 10.1136/adc.2003.037010. PMID 15321956
- [Background] Goncalves-Ferri WA, Martinez FE, Caldas JP, Marba ST, Fekete S, Rugolo L, Tanuri C, Leone C, Sancho GA, Almeida MF, Guinsburg R. Application of continuous positive airway pressure in the delivery room: a multicenter randomized clinical trial. Braz J Med Biol Res. 2014 Feb;47(3):259-64. doi: 10.1590/1414-431X20133278. Epub 2014 Jan 29. PMID 24554040
- [Background] Chernick V, Avery ME. Response of premature infants with periodic breathing to ventilatory stimuli. J Appl Physiol. 1966 Mar;21(2):434-40. doi: 10.1152/jappl.1966.21.2.434. No abstract available. PMID 5949048
- [Background] Dolfin T, Duffty P, Wilkes D, England S, Bryan H. Effects of a face mask and pneumotachograph on breathing in sleeping infants. Am Rev Respir Dis. 1983 Dec;128(6):977-9. doi: 10.1164/arrd.1983.128.6.977. PMID 6650989
- [Background] Fleming PJ, Levine MR, Goncalves A. Changes in respiratory pattern resulting from the use of a facemask to record respiration in newborn infants. Pediatr Res. 1982 Dec;16(12):1031-4. doi: 10.1203/00006450-198212000-00013. PMID 7155672
- [Background] Ramet J, Praud JP, D'Allest AM, Dehan M, Gaultier C. Trigeminal airstream stimulation. Maturation-related cardiac and respiratory responses during REM sleep in human infants. Chest. 1990 Jul;98(1):92-6. doi: 10.1378/chest.98.1.92. PMID 2361419
- [Background] van Vonderen JJ, Kleijn TA, Schilleman K, Walther FJ, Hooper SB, te Pas AB. Compressive force applied to a manikin's head during mask ventilation. Arch Dis Child Fetal Neonatal Ed. 2012 Jul;97(4):F254-8. doi: 10.1136/archdischild-2011-300336. Epub 2011 Dec 5. PMID 22147285